CLINICAL TRIAL: NCT05398939
Title: Impact of COVID-19 Vaccination on Serum 25-hydroxyvitamin D Level
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202204118RINC
Record Dates: First submitted 2022-05-31; First posted 2022-06-01 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-04

CONDITIONS: Acne Vulgaris; Vitamin D Deficiency; COVID-19
MeSH Terms: conditions — Acne Vulgaris; Vitamin D Deficiency; COVID-19 | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acne cohort: Adults with acne vulgaris who are going to receive the third dose of COVID-19 vaccine.
  Interventions: Diagnostic Test: Blood test and skin evaluation

INTERVENTIONS:
Diagnostic Test: Blood test and skin evaluation — The patients received blood tests for serum 25-hydroxyvitamin D level and skin evaluation for severity of acne vulgaris and lesion counts.

SUMMARY:
Vitamin D plays a pivotal but still not well understood role in the immune response to coronavirus disease (COVID-19) infection and vaccination. Many studies also showed a high negative correlation between the severity of inflammatory disease and serum 25-hydroxyvitamin D levels. Patients with acne vulgaris often had deteriorated skin condition after COVID-19 vaccination. Therefore, this study aimed to investigate the relationship of COVID-19 vaccination with serum 25-hydroxyvitamin D level and severity of acne vulgaris.

DETAILED DESCRIPTION:
Vitamin D is known to be related with calcium and bone metabolism. Recently, vitamin D has been shown to play an important role in innate and acquired immunity, cytokine release, inflammatory response, and may be associated with a reduced risk of infection. Studies have reported that serum 25-hydroxyvitamin D concentrations are significantly lower in COVID-19 infected patients than in uninfected patients. In addition, it has been shown that people with higher serum 25-hydroxyvitamin D level would produce significantly more antibodies after COVID-19 vaccination.Thus, it is clear that vitamin D plays a pivotal but still not well understood role in the immune response to COVID-19 infection and vaccination.

Patients with inflammatory skin diseases (e.g., psoriasis, atopic dermatitis, acne vulgaris, hair loss, idiopathic urticaria, etc.) are often observed to have deteriorated skin condition after COVID-19 vaccination, which not only affects the patient's quality of life, but also seriously affects the patient's willingness to complete vaccination. Since many studies have shown a high negative correlation between the severity of inflammatory disease and serum 25-hydroxyvitamin D levels, it is likely that the COVID-19 vaccination also impacts serum 25-hydroxyvitamin D levels. Therefore, this study aimed to analyze the changes in serum 25-hydroxyvitamin D levels and acne severity in patients with acne vulgaris before and after the third dose of COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥ 20 years and < 65 years
2. Diagnosis of acne vulgaris
3. The one will receive the third dose of COVID-19 vaccine
4. Signing informed consent

Exclusion Criteria:

1. History of COVID-19 infection
2. Currently taking vitamin-D, steroid, or any drugs for acne vulgaris.
3. Coagulopathy
4. Having any chronic inflammation disease, immunity-related disease, diabetes, mellitus, kidney disease, or liver disease.
5. Have acute inflammation disease, for example, upper respiratory infection or urinary tract infection
6. Pregnancy or lactation
7. History of cancer or any major systematic disease

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The adults with acne vulgaris who are going to receive the third dose of COVID-19 vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Change in serum 25-hydroxyvitamin D level | 7 days before and 28 days after the third dose of COVID-10 vaccine
  Blood test for serum 25-hydroxyvitamin D level

SECONDARY OUTCOMES:
Change in acne severity | 7 days before and 28 days after the third dose of COVID-10 vaccine
  Skin evaluation by the Global Acne Grading System
Change in acne acne lesion counts | 7 days before and 28 days after the third dose of COVID-10 vaccine
  Counts of acne lesion

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chieh Chan, MD, Principal Investigator — Department of Dermatology, National Taiwan University Hospital
Locations (1):
- Department of Dermatology, National Taiwan University Hospital, Taipei, Taiwan